CLINICAL TRIAL: NCT05367284
Title: Use of Perioperative Testosterone Replacement Therapy (TRT) in Sarcopenic Male Colorectal Cancer Patients - A Single Arm Open Label Feasibility Study
Brief Title: Perioperative Testosterone Replacement Therapy in Sarcopenic Male Colorectal Cancer Patients
Acronym: TERESA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RD21/025
Record Dates: First submitted 2022-01-20; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2021-10

CONDITIONS: Colorectal Cancer; Sarcopenia; Hypogonadism, Male; Perioperative Care; Testosterone Replacement Therapy
MeSH Terms: conditions — Colorectal Neoplasms; Sarcopenia; Eunuchism | interventions — Testosterone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Testosterone — Testogel 16.2 miligrams/ gram (mg/g) gel

SUMMARY:
With increasing age and the additional impact from the bowel cancer and the chemotherapy and/ or radiotherapy it has been described that testosterone (a male hormone produced naturally in the body) levels are reduced. Testosterone has an impact on numerous body functions including the muscle mass and quality. Previous studies have identified that muscle mass is reduced as a result of ageing but also because of the deleterious effect of cancer and chemotherapy and/or radiotherapy. There is growing evidence from published studies that patients with better muscle mass and quality, do better after surgery. Mr Jenkins and his team are therefore looking at ways, the investigators can try and prevent or reduce this muscle loss and therefore improve patient outcomes.

The aim of this study is to assess whether using testosterone replacement therapy in the form of a topically applied gel daily for a total of 12 weeks, is feasible and acceptable by the patients who are diagnosed with colorectal cancer and are waiting to undergo surgery. The investigators will also collect information related to the testosterone replacement therapy such as questionnaires on the quality of life, fatigue and muscle mass, and blood biomarker changes in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 45 years old
* Colorectal cancer - histology confirmed
* Identified as sarcopenic on latest computerised tomography (CT) scan prior to intervention (part of initial investigations - using Martin et al (2013) criteria - 43cm2/m2 for Body Mass Index (BMI) <25, 53cm2/m2 for BMI>25)
* Documented low or normal testosterone at time of recruitment (<12 nano moles/ Litre (nmol/L)
* Eligible for operative intervention
* Capacity to consent
* Able to mobilise & able to complete the 6 Minute Walk Test (MWT)
* Post completion of chemotherapy/ chemoradiotherapy treatment (if the patient has neoadjuvant treatment)
* Booked straight for surgery with an interim of 4-8 weeks.
* Participation in another concurrent trial/ study is accepted, following discussion between the two trial /study teams

Exclusion Criteria:

* Not sarcopenic on computerised tomography (CT)
* Not eligible for surgery
* History of Deep Vein Thrombosis (DVT)/ Pulmonary Embolism (PE)/ prostate cancer/ breast cancer
* Prostate nodule identified during digital rectal examination (DRE) or magnetic resonance imaging (MRI) pelvis
* Multiple distant metastasis which are non-operable
* Prostate specific antigen (PSA) > 3 nanogram/ mililitre (ng/ml)
* Haematocrit (HCT) >52%
* Severe lower urinary tract symptoms
* Class III/ IV heart failure
* Myocardial Infarct or stroke within the last 6 months
* Dementia / No capacity to consent
* Patient on medications with anti-androgen effect eg spironolactone
* Patients with untreated severe obstructive sleep apnoea
* Morbid obesity as defined by Body Mass Index (BMI) >40
* Uncontrolled hypertension
* Patients on long term steroids during the trial period
* Patient on other anabolic agents
* Not already on treatment for primary hypogonadism
* Patients with bone metastasis

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with colorectal cancer who attend to the surgical clinic, following completion of their neoadjuvant chemoradiotherapy or for initial review by the surgical team in order to proceed with surgery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Number of days required for a patient to be recruited on the study and how many patients are recruited | 1 year
  number of days required for patients to be recruited and number of patients recruited by the closure of the study
Number of patients who will complete the 12 week treatment | 12 weeks
  retention of the patients for a the total of 12 weeks by the time of recruitment, will be measured in days on study
Treatment acceptability questionnaire | 12 weeks
  questionnaire on the difficulty experience (Likert scale) for the use of the gel for 12 weeks, if they developed any side effects as described on the CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: JT Jenkins, MD, FRCS, Principal Investigator — London North West University Hospital Healthcare NHS Trust
Locations (1):
- London North West University Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mourtzakis M, Prado CM, Lieffers JR, Reiman T, McCargar LJ, Baracos VE. A practical and precise approach to quantification of body composition in cancer patients using computed tomography images acquired during routine care. Appl Physiol Nutr Metab. 2008 Oct;33(5):997-1006. doi: 10.1139/H08-075. PMID 18923576
- [Background] Mullie L, Afilalo J. CoreSlicer: a web toolkit for analytic morphomics. BMC Med Imaging. 2019 Feb 11;19(1):15. doi: 10.1186/s12880-019-0316-6. PMID 30744586
- [Background] Bozzetti F. Forcing the vicious circle: sarcopenia increases toxicity, decreases response to chemotherapy and worsens with chemotherapy. Ann Oncol. 2017 Sep 1;28(9):2107-2118. doi: 10.1093/annonc/mdx271. PMID 28911059
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Trejo-Avila M, Bozada-Gutierrez K, Valenzuela-Salazar C, Herrera-Esquivel J, Moreno-Portillo M. Sarcopenia predicts worse postoperative outcomes and decreased survival rates in patients with colorectal cancer: a systematic review and meta-analysis. Int J Colorectal Dis. 2021 Jun;36(6):1077-1096. doi: 10.1007/s00384-021-03839-4. Epub 2021 Jan 22. PMID 33481108
- [Background] Lee CM, Kang J. Prognostic impact of myosteatosis in patients with colorectal cancer: a systematic review and meta-analysis. J Cachexia Sarcopenia Muscle. 2020 Oct;11(5):1270-1282. doi: 10.1002/jcsm.12575. Epub 2020 Jun 1. PMID 32483936
- [Background] Pring ET, Malietzis G, Kennedy RH, Athanasiou T, Jenkins JT. Cancer cachexia and myopenia - Update on management strategies and the direction of future research for optimizing body composition in cancer - A narrative review. Cancer Treat Rev. 2018 Nov;70:245-254. doi: 10.1016/j.ctrv.2018.10.002. Epub 2018 Oct 6. PMID 30321741
- [Background] Herbst KL, Bhasin S. Testosterone action on skeletal muscle. Curr Opin Clin Nutr Metab Care. 2004 May;7(3):271-7. doi: 10.1097/00075197-200405000-00006. PMID 15075918
- [Background] Burney BO, Garcia JM. Hypogonadism in male cancer patients. J Cachexia Sarcopenia Muscle. 2012 Sep;3(3):149-55. doi: 10.1007/s13539-012-0065-7. Epub 2012 Apr 20. PMID 22528986
- [Background] Harman SM, Metter EJ, Tobin JD, Pearson J, Blackman MR; Baltimore Longitudinal Study of Aging. Longitudinal effects of aging on serum total and free testosterone levels in healthy men. Baltimore Longitudinal Study of Aging. J Clin Endocrinol Metab. 2001 Feb;86(2):724-31. doi: 10.1210/jcem.86.2.7219. PMID 11158037
- [Background] Feldman HA, Longcope C, Derby CA, Johannes CB, Araujo AB, Coviello AD, Bremner WJ, McKinlay JB. Age trends in the level of serum testosterone and other hormones in middle-aged men: longitudinal results from the Massachusetts male aging study. J Clin Endocrinol Metab. 2002 Feb;87(2):589-98. doi: 10.1210/jcem.87.2.8201. PMID 11836290
- [Background] Slattery ML, Sweeney C, Murtaugh M, Ma KN, Wolff RK, Potter JD, Caan BJ, Samowitz W. Associations between ERalpha, ERbeta, and AR genotypes and colon and rectal cancer. Cancer Epidemiol Biomarkers Prev. 2005 Dec;14(12):2936-42. doi: 10.1158/1055-9965.EPI-05-0514. PMID 16365013
- [Background] Lu Y, Ljung R, Martling A, Lindblad M. Risk of Colorectal Cancer by Subsite in a Swedish Prostate Cancer Cohort. Cancer Control. 2015 Apr;22(2):263-70. doi: 10.1177/107327481502200222. PMID 26068776
- [Background] Gillessen S, Templeton A, Marra G, Kuo YF, Valtorta E, Shahinian VB. Risk of colorectal cancer in men on long-term androgen deprivation therapy for prostate cancer. J Natl Cancer Inst. 2010 Dec 1;102(23):1760-70. doi: 10.1093/jnci/djq419. Epub 2010 Nov 10. PMID 21068432
- [Background] Sah BK, Chen MM, Peng YB, Feng XJ, Yan M, Liu BY, Fan QS, Zhu ZG. Does testosterone prevent early postoperative complications after gastrointestinal surgery? World J Gastroenterol. 2009 Nov 28;15(44):5604-9. doi: 10.3748/wjg.15.5604. PMID 19938202
- [Background] Bhasin S, Storer TW, Berman N, Callegari C, Clevenger B, Phillips J, Bunnell TJ, Tricker R, Shirazi A, Casaburi R. The effects of supraphysiologic doses of testosterone on muscle size and strength in normal men. N Engl J Med. 1996 Jul 4;335(1):1-7. doi: 10.1056/NEJM199607043350101. PMID 8637535
- [Background] Wright TJ, Dillon EL, Durham WJ, Chamberlain A, Randolph KM, Danesi C, Horstman AM, Gilkison CR, Willis M, Richardson G, Hatch SS, Jupiter DC, McCammon S, Urban RJ, Sheffield-Moore M. A randomized trial of adjunct testosterone for cancer-related muscle loss in men and women. J Cachexia Sarcopenia Muscle. 2018 Jun;9(3):482-496. doi: 10.1002/jcsm.12295. Epub 2018 Apr 14. PMID 29654645
- [Background] Walsh JS, Marshall H, Smith IL, Greenfield DM, Swain J, Best E, Ashton J, Brown JM, Huddart R, Coleman RE, Snowden JA, Ross RJ. Testosterone replacement in young male cancer survivors: A 6-month double-blind randomised placebo-controlled trial. PLoS Med. 2019 Nov 12;16(11):e1002960. doi: 10.1371/journal.pmed.1002960. eCollection 2019 Nov. PMID 31714912
- [Background] Wynter-Blyth V, Moorthy K. Prehabilitation: preparing patients for surgery. BMJ. 2017 Aug 8;358:j3702. doi: 10.1136/bmj.j3702. No abstract available. PMID 28790033
- [Background] Santa Mina D, van Rooijen SJ, Minnella EM, Alibhai SMH, Brahmbhatt P, Dalton SO, Gillis C, Grocott MPW, Howell D, Randall IM, Sabiston CM, Silver JK, Slooter G, West M, Jack S, Carli F. Multiphasic Prehabilitation Across the Cancer Continuum: A Narrative Review and Conceptual Framework. Front Oncol. 2021 Jan 11;10:598425. doi: 10.3389/fonc.2020.598425. eCollection 2020. PMID 33505914
- [Background] Jang MK, Park C, Hong S, Li H, Rhee E, Doorenbos AZ. Skeletal Muscle Mass Change During Chemotherapy: A Systematic Review and Meta-analysis. Anticancer Res. 2020 May;40(5):2409-2418. doi: 10.21873/anticanres.14210. PMID 32366384
- [Background] Blauwhoff-Buskermolen S, Versteeg KS, de van der Schueren MA, den Braver NR, Berkhof J, Langius JA, Verheul HM. Loss of Muscle Mass During Chemotherapy Is Predictive for Poor Survival of Patients With Metastatic Colorectal Cancer. J Clin Oncol. 2016 Apr 20;34(12):1339-44. doi: 10.1200/JCO.2015.63.6043. Epub 2016 Feb 22. PMID 26903572
- [Background] Dobs AS, Boccia RV, Croot CC, Gabrail NY, Dalton JT, Hancock ML, Johnston MA, Steiner MS. Effects of enobosarm on muscle wasting and physical function in patients with cancer: a double-blind, randomised controlled phase 2 trial. Lancet Oncol. 2013 Apr;14(4):335-45. doi: 10.1016/S1470-2045(13)70055-X. Epub 2013 Mar 14. PMID 23499390
- [Background] Wu B, Lorezanza D, Badash I, Berger M, Lane C, Sum JC, Hatch GF 3rd, Schroeder ET. Perioperative Testosterone Supplementation Increases Lean Mass in Healthy Men Undergoing Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial. Orthop J Sports Med. 2017 Aug 9;5(8):2325967117722794. doi: 10.1177/2325967117722794. eCollection 2017 Aug. PMID 28840147
- [Background] Shafqat A, Einhorn LH, Hanna N, Sledge GW, Hanna A, Juliar BE, Monahan P, Bhatia S. Screening studies for fatigue and laboratory correlates in cancer patients undergoing treatment. Ann Oncol. 2005 Sep;16(9):1545-50. doi: 10.1093/annonc/mdi267. Epub 2005 May 26. PMID 15919683
- [Background] Del Fabbro E, Garcia JM, Dev R, Hui D, Williams J, Engineer D, Palmer JL, Schover L, Bruera E. Testosterone replacement for fatigue in hypogonadal ambulatory males with advanced cancer: a preliminary double-blind placebo-controlled trial. Support Care Cancer. 2013 Sep;21(9):2599-607. doi: 10.1007/s00520-013-1832-5. Epub 2013 May 8. PMID 23653013
- [Background] Wischmeyer PE, Suman OE, Kozar R, Wolf SE, Molinger J, Pastva AM. Role of anabolic testosterone agents and structured exercise to promote recovery in ICU survivors. Curr Opin Crit Care. 2020 Oct;26(5):508-515. doi: 10.1097/MCC.0000000000000757. PMID 32773614